CLINICAL TRIAL: NCT01512082
Title: The Effect of Pulsed Electromagnetic Field Therapy in Reducing Delayed Onset Muscle Soreness in Marathon Runners. A Double-blind Randomized Placebo-controlled Study.
Brief Title: The Effect of Reducing Soreness in Marathon Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: N-20110021
Record Dates: First submitted 2012-01-10; First posted 2012-01-19 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Contracture of Muscle, Thigh
Keywords: Pain; Delayed onset muscle soreness; Pulsed electromagnetic field; Marathon
MeSH Terms: conditions — Contracture; Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active pulsed electromagnetic field (Experimental)
  Interventions: Device: Pulsed electromagnetic field devices
- Non-active pulsed electromagnetic field (Sham Comparator)
  Interventions: Device: Pulsed electromagnetic field devices

INTERVENTIONS:
Device: Pulsed electromagnetic field devices — Every person received two active devices. The devices emitted 2-ms bursts of 27.12 MHz sinusoidal waves repeating at 2 bursts/s. Peak magnetic field intensity was 0.05 G which induced an average electric field of 10 mV in the tissue with an effect of 7.3 mW/cm3.
  Other Names: ActiPatch TM, Scandinavia ApS, Denmark
  Arms: Active pulsed electromagnetic field
Device: Pulsed electromagnetic field devices — Every persons received two sham pulsed electromagnetic field devices.
  Other Names: ActiPatch TM, Scandinavia ApS, Denmark
  Arms: Non-active pulsed electromagnetic field

SUMMARY:
Delayed onset muscle soreness is defined as the sensition of pain and discomfort in skeletal muscles that occurs after eccentric muscle actions or strenuous exercise like a marathon.

DETAILED DESCRIPTION:
There is a growing body of clinical evidence which shows that noninvasive, nonpharmacologic pulsed electromagnetic fields have many clinical effects. Pulsed electromagnetic fields have shown to reduce pain in different groups of patients. This concerns patients with osteoarthritis, rheumatoid arthritis, diabetic neuropathy, fibromyalgia, distal radius fractures, pelvic pain and postoperative patients.

A marathon is a muscular strain. Physiologic effects of a marathon involves muscular and connective tissue damage which initiates an inflammatory response as well as release of metabolic factors like lactate and free radicals, intracellular metabolites and by-products of proteolysis.

The objective of this study was to investigate the efficacy of pulsed electromagnetic fields compared to placebo in reducing delayed onset muscle soreness in marathon runners.

ELIGIBILITY:
Inclusion Criteria:

* Completion of a marathon
* Age > 18 years

Exclusion Criteria:

- Unable to read and speak Danish

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2011-08; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
Thigh pain by walking | 5 days
  Primary outcome of thigh pain during semi-squat during 5 days following the marathon showed a significantly lower pain among the active group compared to the placebo group.
  The outcome was thigh muscle pain measured on a 10 cm visual analog scale during a squat of 90 degrees three times a day; when they woke up, at 12 pm and 8 pm.

SECONDARY OUTCOMES:
Registration of injuries and symptoms from the musculoskeletal system. | 5 days
  The group that received active pulsed electromagnetic field was running for a significant longer time the first day following the marathon.

CONTACTS AND LOCATIONS:
Overall Officials: Sten Rasmussen, M.D., Principal Investigator — Northern Orthopaedic Division, Aalborg University Hospital, Denmark
Locations (1):
- Orthopaedic Surgery Research Unit, Aalborg University Hospital, Aalborg, Denmark